CLINICAL TRIAL: NCT05535894
Title: Endoscopic Ultrasound-guided Radiofrequency Ablation of Celiac Ganglion for Pain Management and Improvement of Quality of Life in Patients With Unresectable Pancreatic Cancer
Brief Title: Endoscopic Radiofrequency Ablation of Celiac Ganglion for Pain Management and Improvement of Quality of Life in Patients With Unresectable Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Shailendra Singh, Associate Professor & Director, Bariatric Endoscopy, West Virginia University
Other Study IDs: 2202520088
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unresectable Pancreatic Cancer: Endoscopic Ultrasound-guided Radiofrequency Ablation of Celiac Ganglion
  Interventions: Procedure: Ablation of Celiac Ganglion

INTERVENTIONS:
Procedure: Ablation of Celiac Ganglion — Endoscopic Ultrasound-guided Radiofrequency Ablation of Celiac Ganglion

SUMMARY:
This study aims to evaluate the EUS-RFA in terms of efficacy for pain management and improvement in quality-of-life parameters for patients with advanced inoperable pancreatic cancer. The primary objectives of this study are to 1) evaluate the utility of EUS-RFA for pain control and improvement in quality-of-life parameters for patients with advanced pancreatic cancer; 2) to measure the reduction of analgesic medications' requirements in patients affected by inoperable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pancreatic cancer based on clinical, radiological, or pathological assessment;
* Referred for abdominal and/or back pain due to pancreatic cancer;
* No prior history of RFA;
* Cancer pain unresponsive to the WHO 3-step analgesic ladder;
* Willingness to consent to participate in the study.

Exclusion Criteria:

* Patients who are not willing to give informed consent or agree to participate in the study
* Surgically resectable pancreatic cancer;
* Abdominal pain with etiology other than pancreatic malignancy;
* Evidence of concurrent infection;
* Patients with irreversible coagulopathy international normalized ratio >1.5 or platelet count <50,000/mm3),
* Patients with a preliminary diagnosis of adenocarcinoma are not possible established with intraprocedural at EUS-guided FNA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced pancreatic cancer who are deemed as non-surgical candidates
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain severity-BPI | From Baseline up to 3 Months
  Change in severity of pain will be assessed using a standardized the Brief Pain Inventory-Short Form (BPI) ranging from 0 (no pain) to 10 (worst pain possible).
Pain severity-VAS | From Baseline up to 3 Months
  Change in severity of pain will be assessed using visual analog scale (VAS) ranging from 0 (no pain) to 10 (worst pain possible).
Pain severity-NRS | From Baseline up to 3 Months
  Change in severity of pain will be assessed using numerical rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain possible).
Quality of Life (EORTC PAN26) | From Baseline up to 3 Months
  Changes in Quality of Life as scored with the Europen Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire pancreatic cancer module (PAN26). This measure uses a Likert type scale 1-4 with 1=better and 4=worse.
Quality of Life (EORTC C30) | From Baseline up to 3 Months
  Changes in Quality of Life as scored with the EORTC Quality of Life Questionnaire core questionnaire (C30). This measure uses a Likert type scale 1-4 with 1=better and 4=worse.
Quality of Life (NFHSI) | From Baseline up to 3 Months
  Changes in Quality of Life as scored with the National Comprehensive Cancer Network Functional Assessment of Cancer Therapy Hepatobiliary-Pancreatic Symptom Index (NFHSI). This measure uses a Likert type scale 0-4 with 0=no symptoms and 4= worst symptoms.
Concomitant Analgesic/Narcotic Use | From Baseline up to 3 Months
  Percent change in concomitant analgesic therapy will be evaluated. Details on the dose and frequency of opioid medications administered within 24 hours before the intervention will be collected and at different follow-up intervals after the procedure. The total dose of analgesic therapy administered will then be converted into an oral morphine equivalent dose for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Shailendra Singh, MD, Principal Investigator — West Virginia University
Locations (1):
- Shailendra Singh, Morgantown, West Virginia, United States